CLINICAL TRIAL: NCT00030342
Title: A Phase I/II Study Of Interleukin-12-Primed Activated T Cells In Combination With 5FU, GM-CSF And Interferon Alfa-2b In Metastatic Renal Cell Carcinoma Or Colorectal Carcinoma
Brief Title: Biological Therapy and Chemotherapy in Treating Patients With Metastatic Kidney Cancer or Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Luke's Medical Center (Other)
Responsible Party: John P. Hanson, Jr, Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: STLMC-IMM-0104; CDR0000069153 (Registry Identifier: PDQ (Physician Data Query)); STLMC-L-01108; NCI-V01-1686
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2008-10

CONDITIONS: Colorectal Cancer; Kidney Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Colorectal Neoplasms; Kidney Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; sargramostim; Fluorouracil

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: sargramostim
Biological: therapeutic autologous lymphocytes
Drug: fluorouracil

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining biological therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of biological therapy combined with chemotherapy in treating patients who have metastatic kidney cancer or colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of a repeat course of interleukin-12-primed activated T cells (12ATC) in combination with fluorouracil, sargramostim (GM-CSF), and interferon alfa-2b in patients with metastatic renal cell or colorectal carcinoma.
* Determine the clinical responses of patients treated with this regimen.
* Determine the efficacy of 12ATC in these patients.
* Determine whether there are changes in immunologic parameters related to 12ATC as measured by lymphocyte phenotype and cytokine secretion in these patients.
* Determine the correlation between clinical responses in patients treated with this regimen and in vitro immune functions of lymphocytes.

OUTLINE: Patients are stratified according to disease type (renal cell carcinoma vs colorectal carcinoma).

Patients receive sargramostim (GM-CSF) subcutaneously (SC) daily on days 1-5 and then undergo collection of autologous peripheral blood mononuclear cells (PBMC) on days 6 and 7 of week 1. The PBMC are treated ex vivo to form interleukin-12-primed activated T cells (12ATC).

Patients receive fluorouracil IV over 24 hours on day 6 of week 2 and interferon alfa-2b SC and GM-CSF SC 3 times weekly on weeks 3-5. Patients receive 12ATC IV over 15-30 minutes twice weekly and interferon alfa-2b SC (at least 24 hours after 12ATC infusion) once weekly on weeks 6-8. Patients with complete or partial response or stable disease at 3 weeks after the last 12ATC infusion may receive an additional 8-week course as above.

Patients are followed every 2-3 months for 1 year and then every 6 months for 2 years or at any time when the physical examination or symptoms are suspicious for tumor progression.

PROJECTED ACCRUAL: A total of 60 patients (30 per stratum) will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic renal cell carcinoma or colorectal carcinoma, meeting 1 of the following criteria:

  * Obtained no benefit from prior standard or salvage therapy
  * Ineligible for standard therapy because of concurrent illness
  * Declined standard therapy
* At least 1 site of measurable disease that can be measured in at least 1 dimension

  * At least 20 mm with conventional techniques OR at least 10 mm with spiral CT scan
* No untreated or unstable, treated brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 4,000/mm^3
* Granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* No coagulation disorders

Hepatic:

* Bilirubin no greater than 2.5 mg/dL*
* ALT/AST less than 3 times upper limit of normal*
* PT no greater than 1.5 times control (unless therapeutically anticoagulated)
* PTT less than 1.5 times control (unless therapeutically anticoagulated) NOTE: *Patients whose cancer has led to values that do not fall within the above ranges may be eligible at the discretion of the investigators

Renal:

* Creatinine no greater than 2.0 mg/dL* NOTE: *Patients whose cancer has led to values that do not fall within the above range may be eligible at the discretion of the investigators

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No thrombophlebitis

Pulmonary:

* FEV_1 and FVC at least 65% predicted
* No uncontrolled pulmonary embolism

Other:

* No other malignancy within the past 5 years except resected basal cell skin cancer or carcinoma in situ of the cervix
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to interleukin-12-primed activated T cells or other study agents
* No active autoimmune disease
* No uncontrolled thyroid abnormalities
* No ongoing or active infection
* No other uncontrolled concurrent illness
* No psychiatric illness or social situations that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 2 years after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 4 weeks since prior immunotherapy

Chemotherapy:

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* At least 4 weeks since prior steroid therapy or steroid-containing compounds
* At least 2 weeks since prior topical or inhaled steroids

Radiotherapy:

* More than 4 weeks since prior radiotherapy and recovered

Surgery:

* More than 4 weeks since prior major surgery

Other:

* No other concurrent investigational agents
* No other concurrent commercial anticancer agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2001-11; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Response as measured by RECIST guidelines and Kaplan-Meier method at 5 years
Survival as measured by the Kaplan-Meier method at 5 years
Safety as measured by NCI common toxicity table at study completion

CONTACTS AND LOCATIONS:
Overall Officials: John P. Hanson, MD, Study Chair — St. Luke's Medical Center
Locations (1):
- Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin, United States